## The Effect of Structured Reminiscence on the Symptom Management, Life Satisfaction, and Self-Transcendence of Palliative Care Patients: A Randomized Placebo-Controlled Trial



Fig. 1. CONSORT flow chart

## **TABLES**

Table 1. Distribution of patients' sociodemographic and disease-related characteristics

| Variables | Total<br>n=44 | Interventio<br>n<br>n=15 | Placebo<br>n=14 | Control<br>n=15 | р |
|---|---|---|---|---|---|
| Age (years), Mean ± SD | 64.93 ± 3.69 | 65.67 ± 3.67 | 64.57 ± 4.15 | 65.60 ± 2.56 | ~-0 CEE 3 |
| %95 CI | 64.24, 66.35 | 63.63, 67.70 | 62.18, 66.97 | 64.18, 67.02 | p=0.655 ° |
| Age Groups, n (%) | | | | | |
| < 65 years | 13 (29.5) | 4 (26.7) | 4 (28.6) | 5 (33.3) | p=0.844 b |
| ≥ 65 years | 31 (70.5) | 11 (73.3) | 10 (71.4) | 10 (66.7) | |
| Gender, n (%) | | | | | |
| Female | 17 (38.6) | 5 (33.3) | 6 (42.9) | 6 (40.0) | p=0.853 b |
| Male | 27 (61.4) | 10 (66.7) | 8 (57.1) | 9 (60.0) | |
| Marital status, n (%) | | | | | |
| Married | 38 (86.4) | 14 (93.3) | 11 (78.6) | 13 (86.7) | p=0.796 b |
| Single/widowed/divorced | 6 (13.6) | 1 (6.7) | 3 (21.4) | 2 (13.3) | |
| Primer Disease, n (%) | , , | , , | , , | , , | |
| Cancer | 31 (70.5) | 10 (66.7) | 11 (78.6) | 10 (66.7) | |
| Cardiovascular System | 5 (11.4) | 2 (13.3) | 1 (7.1) | 2 (13.3) | 0 000 c |
| Neurological System | 3 (6.8) | 2 (13.3) | 1 (7.1) | ` | p=0.829 <sup>c</sup> |
| Respiratory System | 3 (6.8) | | 1 (7.1) | 2 (13.3) | |
| Urinary System | 2 (4.5) | 1 (6.7) | | 1 (6.7) | |
| Cancer Localization (n=31), n(%) | , , | , , | | , , | |
| Genitourinary | 8 (25.8) | 2 (20) | 3 (27.3) | 3 (30.0) | |
| Respiratory | 7 (22.6) | 3 (30) | 2 (18.2) | 2 (20.0) | 0.047 h |
| Gastrointestinal | 7 (22.6) | 2 (20) | 2 (18.2) | 3 (30.0) | p=0.817 b |
| Breast | 5 (16.2) | 2 (20) | 2 (18.2) | 1 (10.0) | |
| Hematological | 4 (12.9) | 1 (10) | 2 (18.2) | 1 (10.0) | |
| Duration of the disease (years) | | | | | |
| Mean ± SD | | | 5.71 ± 2.97 | | p=0.465 a |
| 95% CI | 4.12, 6.15 | 3.37, 5.17 | 4.00, 7.43 | 2.85, 8.08 | • |
| Length of stay in the unit | | | | | |
| <1 week | 34 (77.2) | 11 (73.4) | 11 (78.6) | 12 (80.0) | |
| 1- 2 weeks | 5 (11.4) | 2 (13.3) | 1 (7.1) | 2 (13.3) | p=0.936 b |
| >2 weeks | 5 (11.4) | 2 (13.3) | 2 (14.3) | 1 (6.7) | p=0.930 ° |
| ECOG Performance Scale | 4 (0.4) | 1 (0.7) | 4 (7 4) | 0 (40 0) | |
| 1 | 4 (9.1) | 1 (6.7) | 1 (7.1) | , , | |
| 2 | 7 (15.9) | 2 (13.3) | 3 (21.4) | 2 (13.3) | p=0.955 b |
| 3 | 28 (63.6) | 10 (66.7) | 8 (57.1) | 10 (66.7) | |
| 4 | 5 (11.4) | 2 (13.3) | 2 (14.3) | 1 (6.7) | |

SD: Standard Deviation; CI: confidence interval; a One Way ANOVA; b Chi-square test; c Fisher's exact test

Table 2. Comparison of the symptom assessment sub-scale and total score averages of the groups within and between groups

| | Groups | Intervention | Placebo | Control | | |
|---|---|---|---|---|---|---|
| | | n=15 | n=14 | n=15 | $X^2$ | р |
| | | Mean ± SD | Mean <b>±</b> SD | Mean <b>±</b> SD | | |
| _ | Pre-test | 1.58 ± 0.56 | 1.49 ± 0.32 | 1.52 ± 0.29 | 0.218 | 0.897 |
| ဟ် <u> </u> | Post-test | 1.46 ± 0.50 | $1.45 \pm 0.27$ | 1.50 ± 0.28 | 0.461 | 0.794 |
| SASM Solution SASM Solution Sample Sa | | -2.718 | -2.379 | -1.841 | | |
| ž | р | 0.007* | 0.017* | 0.066 | | |
| | Δ | - 7.60% | - 2.68% | - 1.31% | | |
| | Pre-test | 1.40 ± 0.65 | 1.41 ± 0.68 | 1.41 ± 0.63 | 0.097 | 0.953 |
| S-<br>cal | Post-test | 1.43 ± 0.62 | | | 0.356 | 0.837 |
| MSAS-<br>Physica | Z | -1.099 | -0.730 | -0.942 | | |
| WSAS-<br>Physical Z<br>p | | 0.272 | 0.465 | 0.346 | | |
| _ | Δ | + 2.14% | - 0.71% | 0% | | |
| | Pre-test | 1.18 ± 0.70 | 1.29 ± 0.62 | 1.28 ± 0.59 | 0.556 | 0.757 |
| S-<br>Po | Post-test | $0.91 \pm 0.46$ | 1.11 ± 0.48 | 1.32 ± 0.58 5.36 | | 0.068 |
| MSAS-<br>Psycho | Z | -2.977 | -2.695 | -1.705 | | |
| -SASA Post-test Z p | | 0.003* | 0.007* | 0.088 | | |
| | Δ | - 22.88% | - 13.95% | + 3.13% | | |
| | Pre-test | 1.07 ± 0.48 | 1.13 ± 0.47 | 1.10 ± 0.44 | 0.715 | 0.699 |
| MSAS-<br>Total | Post-test | 1.06 ± 0.45 | 1.12 ± 0.47 | 1.11 ± 0.43 | 0.246 | 0.884 |
| | Z | -0.881 | -1.468 | -0.395 | | |
| | р | 0.378 | 0.142 | 0.693 | | |
| | <u> </u> | - 0.93% | - 0.88% | + 0.91% | | |

MSAS: Memorial Symptom Assessment Scale; SD: Standard Deviation; Δ: percentage of change; Z: Wilcoxon signed-ranks test; X<sup>2</sup>: Kruskal Wallis H test; \*p<0.05; \*\*p<0.001

Table 3. Comparison of the mean scores of the groups on the life satisfaction scores within and between groups

| | Contentment With Life Assessment Scale | | | | |
|---|---|---|---|---|---|
| | Pre-test | Post-test | Δ | t | р |
| | Mean ± SD | Mean ± SD | | | · |
| Intervention (n=15) | 16.27 ± 2.68 | 21.66 ± 2.37 | + 33.12% | -7.155 | <0.001** |
| Placebo (n=14) <sup>2</sup> | 16.14 ± 2.31 | 17.21 ± 2.15 | + 6.63% | -2.206 | 0.046* |
| Control (n=15) 3 | 16.20 ± 2.35 | 15.40 ± 1.91 | - 4.93% | 1.922 | 0.075 |
| F | 0.031 | 16.817 | | | |
| р | 0.990 | <0.001** | | | |
| Post-hoc | | 1>2,3 | | | |
| | Gro | up Time Interacti | ion | | |
| | Group | Time | Group*Time | | |
| $F_2$ | 6.342 | 32.376 | 31.195 | | |
| р | 0.004* | <0.001** | <0.001** | | |
| η² | 0.236 | 0.441 | 0.603 | | |
| Post-hoc | | 1>2,3 | | | |
| | Pi | re-test < Post-tes | st | | |

SD: Standard Deviation;  $\Delta$ : percentage of change; t: Paired-samples t test; F: One Way ANOVA; F<sub>2</sub>: Repeated measures ANOVA;  $\eta^2$ : Eta-square; \*p<0.05; \*\*p<0.001

Table 4. Comparison of the self-transcendence mean scores of the groups within and between groups

| | | Pre-test<br>Mean <b>±</b> SD | Post-test<br>Mean <b>±</b> SD | Δ | | t | р |
|---|---|---|---|---|---|---|---|
| Intervention (n=15 | ) 1 | 35.80 ± 4.36 | 43.93 ± 5.39 | + 22. | 71% | -14.321 | <0.001* |
| Placebo (n=14) <sup>2</sup> | | 36.28 ± 5.10 | 38.50 ± 6.00 | + 6.1 | 2% | -2.090 | 0.057 |
| Control (n=15) <sup>3</sup> | | 35.53 ± 4.94 | 35.60 ± 5.86 | + 0.2 | 20% | -0.065 | 0.949 |
| | F | 0.244 | 10.312 | | | | |
| | р | 0.784 | <0.001** | | | | |
| Pos | t-hoc | | 1>2,3 | | | | |
| | | Group Time | Interaction | | | | |
| | Group | Tim | e Grou | up*Time | | | |
| F <sub>2</sub> | 4.177 | 43.8 | 70 2 | 1.616 | | | |
| р | 0.022 | * <0.00 | )1** <0 | .001** | | | |
| η² | 0.169 | 0.51 | 17 0 | .513 | | | |
| Post-hoc | | 1>2 | 2,3 | | | | |
| | | Pre-test < | Post-test | | | | |

 $\begin{tabular}{lll} \hline Pre-test &< Post-test \\ \hline \hline SD: Standard Deviation; $\Delta$: percentage of change; t: Paired-samples t test; $F$: One Way ANOVA; $F_2$: Repeated measures ANOVA; $\eta^2$: Eta-square; *p<0.05; **p<0.001 \\ \hline \end{tabular}$